CLINICAL TRIAL: NCT03190850
Title: Effect of Inspiratory Muscle Training in Sleep Apnea of Elderly
Brief Title: Effect of Inspiratory Muscle Training
Acronym: MARITSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150276
Record Dates: First submitted 2017-03-23; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea; Elderly; Inspiratory training
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator will not know the final result of the tests performed until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention: Exercises wih load Device: "Powerbreathe"
  Interventions: Other: Intervention
- Control (Placebo Comparator): Control: Exercises without load
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — The device in which the breathing exercises will be performed will be adjusted with progressive loading aiming to improve muscular strength
  Arms: Intervention
Other: Control — The device in which the breathing exercises will be performed will not be adjusted with progressive loading.
  Arms: Control

SUMMARY:
This study aims to evaluate the effect of inspiratory muscle training on sleep apnea in the elderly. The patients screened will be randomized and allocated into two groups, intervention and control. In the intervention group, the patients will perform the exercises with the inspiratory muscular training apparatus called Powerbreathe with progressive load, according to its inspiratory muscular force. The control group will perform the same exercises, with the same apparatus, but without load.

DETAILED DESCRIPTION:
At the beginning of the study the patients will be evaluated initially with polysomnography. Patients who meet the inclusion criteria and sign the consent form will be evaluated with the following exams before and after inspiratory muscle training: manovacuometry, spirometry, diaphragmatic ultrasound and an anthropometric evaluation. After inspiratory muscle training, all patients will also perform polysomnography again to check for apnea-hypopnea index change.The patients screened will be randomized and allocated into two groups, intervention and control. In the intervention group, the patients will perform the exercises with the inspiratory muscular training apparatus called Powerbreathe with progressive load, according to its inspiratory muscular force. The control group will perform the same exercises, with the same apparatus, but without load.Patients in the intervention group will perform inspiratory muscle training as follows: in the first and second weeks, the patients will be instructed to perform the breathing exercises three times a week, performing four sets of six repetitions with one minute rest, with load of 50% of the maximum inspiratory pressure that will be preset in the Powerbreathe device by the study collaborators. At the end of the second week, they will perform reassessment of inspiratory pressures (MIP) and maximal expiratory pressure, with a 75% load adjustment of the PIM in the Powerbreathe device, and the patients being instructed to perform the same series and repetitions with frequency of exercise in five times in the week in the third and fourth week. At the end of the fourth week, they will perform a reassessment of the inspiratory pressures (MIP) and maximal expiratory pressures, with a 75% load adjustment of the MIP in the Powerbreathe device and the patients being instructed to perform the same series and repetitions with frequency of exercise in five times in the week on the fifth and sixth week. At the end of the sixth week, they will perform a reassessment of inspiratory pressures (MIP) and maximal expiratory pressure, with a 80% load adjustment of the MIP in the Powerbreathe device and the patients being instructed to perform the same series and repetitions with frequency of exercise in seven times in the week in the seventh and eighth week. The no-load (control) inspiratory muscle training group will perform the same series, repetitions and frequency of breathing exercises and reassessments of the intervention group, but there will be no load adjustment on the Powerbreathe appliances of this group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 80 years
* Both genders
* Not be treating apnea with AHI between 10 and 30
* Do not tolerate or not have access to CPAP with any AHI
* To consent to participate in the research

Exclusion Criteria:

* Treatment for sleep apnea
* Severe chronic illness
* IAH greater than 35
* Uncontrolled arterial hypertension
* Acute myocardial infarction
* Recent upper airway trauma
* High performance athletes
* Medications with effect on the central nervous system

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04-05 (Actual); Primary Completion 2018-03-09 (Estimated); Study Completion 2018-05-10 (Estimated)

PRIMARY OUTCOMES:
Effect of inspiratory exercise on apnea-hypopnea index in elderly patients with sleep apnea. | 8 weeks
  Impact of inspiratory muscle training on apnea-hypopnea index in elderly patients with sleep apnea. The measurement will be taken before and after the training. The measurement is apnea-hypopnea index through polysomnograph

SECONDARY OUTCOMES:
Effect of inspiratory training on maximal inspiratory and expiratory pressures | 8 weeks
  Impact of training muscle inspiratory on muscle strength inspiratory and expiratory measured through manovacuometry. The measurement will be taken before and after the training
Effect of inspiratory muscle training on diaphragm thickness | 8 weeks
  Impact of training muscle inspiratory on diaphragm thickness measured through diaphragmatic ultrasound. The measurement will be taken before and after the training.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Martinez, Study Director — PhD of Graduate Program in Medical Sciences
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided